CLINICAL TRIAL: NCT01656876
Title: The Effects of Mirror Therapy on Upper Extremity in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: CRC-09-10-08
Record Dates: First submitted 2012-07-27; First posted 2012-08-03 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2012-11

CONDITIONS: Cerebrovascular Accident
Keywords: Comparative effectiveness research; Mirror therapy; Stroke rehabilitation; Clinical evaluation; Kinematic analysis; Mesh glove; Combined therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mirror therapy (Experimental): mirror box training with or without sham mesh glove stimulation
  Interventions: Behavioral: Mirror box training
- Mirror therapy + Mesh glove stimulation (Experimental): Mirror therapy combined with mesh glove stimulation
  Interventions: Behavioral: Mirror box training; Other: mesh glove stimulation
- Controlled intervention (Active Comparator): conventional interventions
  Interventions: Behavioral: conventional intervention

INTERVENTIONS:
Behavioral: Mirror box training — This protocol includes 1 hour mirror therapy and 0.5 hour functional training in a session. The treatment intensity is 1.5 hours/day, 5 days/week, for 4 weeks. MT focuses on symmetrical bimanual movements and simultaneously observing the visual feedback of the unaffected upper extremity reflected by the mirror.
  Other Names: MT
  Arms: Mirror therapy; Mirror therapy + Mesh glove stimulation
Other: mesh glove stimulation — The MG is a two-channel electrical stimulator providing synchronous or reciprocal sensory stimulation with variant amplitudes.
  Other Names: MG
  Arms: Mirror therapy + Mesh glove stimulation
Behavioral: conventional intervention — Participants in this group receive a structured protocol based on occupational therapy such as neuro-developmental techniques and task-oriented approach
  Other Names: CI
  Arms: Controlled intervention

SUMMARY:
The purpose of this study is to compare treatment efficacy of mirror therapy (MT), mirror therapy combining mesh glove (MG+MT) stimulation, and controlled treatment (CT) in people with stroke.

DETAILED DESCRIPTION:
55% to 75% of people after stroke have a paretic arm that causes motor impairment. Among novel rehabilitation interventions, MT was found to be beneficial and comparatively low-cost. MT reduced motor impairment possibly in part of recruiting the premotor cortex or balancing the neural activation within the primary motor cortex toward the affected hemisphere. However, the benefits in certain aspects of outcomes are under debate. Another treatment, MG, can be used to normalize muscle tone, suppress muscle spasticity, enhance residual volitional activity of hand and arm, or even increasing walking speed. In addition, providing MG stimulation might result in plastic changes in the primary motor cortex, and induced a long-lasting modulated effect on motor cortical excitability. The possible mechanism of brain plasticity underlying MG is collective with the mechanism behind the MT. Adding MG to MT might augment the cortical reorganization. In sum, combining MT with MG may supplement the disadvantage or uncertain effects of MT and broaden the benefited outcomes.

ELIGIBILITY:
Inclusion Criteria:

* The onset duration more than 3 months
* Demonstration of Brunnstrom stage equal to or above stage III of the affected upper extremity
* No serious cognitive deficits (a score of more than 24 on the Mini Mental State Exam)
* No serious visual and visual-perception impairments
* No concurrent participation in other drug or rehabilitation research
* No serious attention deficits
* No excessive spasticity in any of the joints of the affected UL exclusion criteria

Exclusion Criteria:

* Exhibit physician determined major medical problems or poor physical conditions that would interfere with participation
* Excessive pain in any joint that might limit participation

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment (FMA) | Baseline, change from baseline in FMA at 4 weeks, change from baseline in FMA at 16 weeks, change from baseline in FMA at 28 weeks
  The upper-extremity subscale of the FMA contains 33 items to assess motor impairment. Each item is scored on a 3-point ordinal scale (0-cannot perform, 1-performs partially, 2-performs fully and correctly). The sub-score of a proximal shoulder/elbow (0-42) and a distal hand/wrist (0-24) will be also calculated to investigate the treatment effects on separate upper extremity elements.
Wolf Motor Function Test (WMFT) | Baseline, change from baseline in WMFT at 4 weeks, change from baseline in WMFT at 16 weeks, change from baseline in WMFT at 28 weeks
  * The WMFT composed of 3 parts: Time, Functional ability, and Strength
  * Includes 15 function-based tasks and 2 strength based tasks
  * Performance time is referred to as WMFT-TIME
  * Functional ability is referred to as WMFT-FAS
  * Items 1-6 involve timed functional tasks, items 7-14 are measures of strength, and the remaining 9 items consist of analyzing movement quality when completing various tasks.
  * Examiner should test the less affected upper extremity followed by the most affected side.
  * Uses a 6-point ordinal scale
  * "0" = "does not attempt with the involved arm" to
  * "5" = "arm does participate; movement appears to be normal."
  * Maximum score is 75
  * Lower scores are indicative of lower functioning levels
  * WMFT-TIME allows 120 seconds per task
Accelerometers | Baseline, change from baseline in accelerometers at 4 weeks, change from baseline in accelerometers at 16 weeks, change from baseline in accelerometers at 28 weeks
  The accelerometers are used to provide a direct and objective measure of the amount of the impaired arm movement outside the laboratory. Acceleration is sampled at 10 Hz and summed over a user- specified epoch. The recording epoch in this study is 2 seconds; recording capacity is approximately 72 hours. A "threshold-filter" will be applied to the raw recordings to obtain an accurate measure of the duration of arm movement.
revised Nottingham Sensory Assessment (rNSA) | Baseline, change from baseline in rNSA at 4 weeks, change from baseline in rNSA at 16 weeks, change from baseline in rNSA at 28 weeks
  The rNSA examines the sensory function of the affected arm and includes tactile sensation (0=Absent, 1=Impaired, 2=Normal), proprioception (0=Absent, 1=Appreciation of movement sense, 2=Direction of movement sense, 3=Joint position sense), and stereognosis (0=Absent, 1=Impaired, 2=Normal) subtests.

SECONDARY OUTCOMES:
Kinematic analyses | Baseline, change from baseline in kinematic parameters at 4 weeks
  A 7-camera motion-analysis system (VICON MX, Oxford Metrics Inc., Oxford, UK) was used. The variables of reaction time (second), movement time (second), total displacement (mm), peak velocity (mm/second), percentage of peak velocity, joint recruitments (degree), and maximum shoulder and elbow cross-correlation were collected.
Motor Activity Log (MAL) | Baseline, change from baseline in MAL at 4 weeks, change from baseline in MAL at 16 weeks, change from baseline in MAL at 28 weeks
  The MAL is a semi-structured interview of patients to assess the amount of use (AOU) and quality of movement (QOM) of the affected upper extremity in 30 important daily activities using a 6-point ordinal scale. Higher scores indicate superior amount and quality of use in affected upper extremity.
Semmes-Weinstein monofilaments | Baseline, change from baseline in Semmes-Weistein monofilaments at 4 weeks, change from baseline in Semmes-Weistein monofilaments at 16 weeks, change from baseline in Semmes-Weistein monofilaments at 28 weeks
  The Semmes-Weinstein monofilaments is used for measuring diminishing and returning cutaneous sensation.A nylon 'string' is specifically calibrated in stiffness to represent a baseline level of sensation that can be considered 'the line' between having neuropathy and having normal sensation.
Functional Independence Measure (FIM) | Baseline, change from baseline in FIM at 4 weeks, change from baseline in FIM at 16 weeks, change from baseline in FIM at 28 weeks
  The FIM consists of 18 items grouped into 6 subscales. Each item is rated from 1 to 7 (max. score 126) based on the required level of assistance to perform the tasks.
Stroke Impact Scale version 3.0 (SIS 3.0) | Baseline, change from baseline in SIS at 4 weeks, change from baseline in SIS at 16 weeks, change from baseline in SIS at 28 weeks
  The SIS is a stroke-specific instrument of health related quality of life and contains 59 items measuring 8 domains. Items are rated on a 5- point Likert scale with lower scores indicate greater difficulty in task completion during the past week. Aggregate scores, ranges from 0 to 100, are generated for each domain.
8-OHdG | Baseline, change from baseline in 8-OHDG at 4 weeks, change from baseline in 8-OHDG at 16 weeks, change from baseline in 8-OHDG at 28 weeks
  Urinary 8-OHdG is a stable and integral biomarker of oxidative DNA damage.About 10 mL to 15 mL urine samples of the patients will be collected in the centrifugal tubes before and after rehabilitation interventions. The samples will be transported with dry ice under 4°C and preserved in a -80°C refrigerator before analysis. A highly sensitive and selective method, using isotope- dilution liquid chromatography with tandem mass spectrometry (LC/MS/MS), will be used to determine the urinary 8-OHdG levels.

CONTACTS AND LOCATIONS:
Overall Officials: Tsan-hon Liou, PhD, Principal Investigator — Shuang-Ho Hospital, Taipei Medical University; Ching-yi Wu, ScD, Principal Investigator — Department of Occupational Therapy, College of Medicine, Chang Gung University; Keh-chung Lin, ScD, Principal Investigator — School of Occupational Therapy, College of Medicine, National Taiwan University
Locations (1):
- Shuang-Ho Hospital, Taipei Medical University, New Taipei City, Taiwan